CLINICAL TRIAL: NCT05060627
Title: An Open Label, Multicenter, Phase I/II Study of Belantamab Mafodotin in Combination With Kd for the Treatment of Relapsed Myeloma Patients, Refractory to Lenalidomide.
Brief Title: Study of Belantamab Mafodotin in Combination With Kd for the Treatment of Relapsed Myeloma Patients, Refractory to Lenalidomide
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: PETHEMA Foundation (Other)
Collaborators: Adknoma Health Research (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GEM-BELMA; 2021-002125-15 (EudraCT Number)
Record Dates: First submitted 2021-09-17; First posted 2021-09-29 (Actual); Last update posted 2022-09-08 (Actual); Status verified 2022-09

CONDITIONS: Relapsed Multiple Myeloma
Keywords: Relapsed multiple myeloma; Refractoriness to lenalidomide
MeSH Terms: conditions — Multiple Myeloma | interventions — belantamab mafodotin; carfilzomib; Dexamethasone

STUDY DESIGN:
Intervention Model Description: A phase I classic 3+3 design, to establish the maximum tolerated dose (MTD) of the combination. Once the MTD will be defined, a dose expansion phase II will be open to recruit up to 60 patients.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Belantamab-Mafodotin + Carfilzomib+ dexametasona (Experimental): In the phase 1 of the study, aiming to establish the recommended phase 2 dose (RP2D), patients will be included following the classic 3 + 3 design.
  Once the DLT assessment period is completed and the MTD is defined, the recruitment will continue in the expansion phase 2.
  Combination treatment will be administered at the recommended Phase 2 dose (RP2D) based on the results of the phase 1 dose escalation part of the study:
  * Belantamab mafodotin on day 1 at the RP2D, every 8 weeks, intravenously (IV).
  * Carfilzomib will be given at the RP2D weekly IV on days: 1, 8, and 15 of every 4-week cycle (Q4W).
  * Dexamethasone will be given at the dose of 40 mg (or 20 mg if patient > 75 years old) on days: 1, 8, 15 and 22 Q4W.
  From month 13 onwards carfilzomib treatment will be given on day 1 and 15 of every 4-weeks cycles. Belantamab will be given at the RP2D every 8 weeks and Dexamethasone 40mg on days 1, 8, and 15 of every 4-week cycle.
  Interventions: Drug: Belantamab mafodotin; Drug: Carfilzomib; Drug: Dexamethasone

INTERVENTIONS:
Drug: Belantamab mafodotin — In phase 1:
  * Dose level -1: Belantamab-Mafodotin 1.9 mg/kg day 1, Q8W
  * Dose level 1,2,3: Belantamab-Mafodotin 2.5 mg/kg day 1, Q8W In phase 2: maximum tolerated dose (MTD) of the combination
Drug: Carfilzomib — In phase 1:
  * Dose level -1, 1: Carfilzomib 20/45 mg/m2 days 1, 8, and 15, Q4W.
  * Dose level 2: Carfilzomib 20/56 mg/m2 on days 1, 8, and 15, Q4W
  * Dose level 3: Carfilzomib 20/70 mg/m2 on days 1, 8, and 15, Q4W.
  In phase 2: maximum tolerated dose (MTD) of the combination
Drug: Dexamethasone — Description: Dexamethasone 40 mg weekly (days 1, 8, 15 and 22) or 20 mg in patients > 75 years old., Q4W

SUMMARY:
This is a phase I-II open-label, multicenter, non-randomized study aiming to evaluate the efficacy and safety of belantamab mafodotin in combination with carfilzomib (Kyprolis®) and dexamethasone (Kd). Since this is the first time that this combination is being evaluated in a clinical trial, a first dose escalation part will be developed following the classic 3+3 design, to establish the maximum tolerated dose (MTD) of the combination. Once the MTD will be defined, a dose expansion phase will be open to recruit up to 60 patients.

Patients will receive treatment with belantamab-mafodotin + Kd, until unacceptable toxicity, disease progression, patient withdrawal, loss to follow-up, end of study, or death.

DETAILED DESCRIPTION:
This is a phase I-II open-label, multicenter, non-randomized study aiming to evaluate the efficacy and safety of belantamab mafodotin in combination with carfilzomib (Kyprolis®) and dexamethasone (Kd). Since this is the first time that this combination is being evaluated in a clinical trial, a first dose escalation part will be developed following the classic 3+3 design, to establish the maximum tolerated dose (MTD) of the combination. Once the MTD will be defined, a dose expansion phase will be open to recruit up to 60 patients.

The study comprises the following phases:

Phase 1 (Lead-in): 3+3 Dose escalation

In the phase 1 of the study, aiming to establish the recommended phase 2 dose (RP2D), patients will be included following the classic 3 + 3 design. Dose levels will be as follows:

Dose level -1

* Belantamab-Mafodotin 1.9 mg/kg day 1, Q8W
* Carfilzomib 20/45 mg/m2 on days 1, 8, and 15, Q4W.
* Dexamethasone 40 mg weekly (days 1, 8, 15 and 22) or 20 mg in patients > 75 years old, Q4W Dose level 1
* Belantamab-Mafodotin 2.5 mg/kg day 1, Q8W
* Carfilzomib 20/45 mg/m2 days 1, 8, and 15, Q4W.
* Dexamethasone 40 mg weekly (days 1, 8, 15 and 22) or 20 mg in patients > 75 years old., Q4W Dose level 2
* Belantamab-Mafodotin 2.5 mg/kg on day 1, Q8W
* Carfilzomib 20/56 mg/m2 on days 1, 8, and 15, Q4W.
* Dexamethasone 40 mg weekly (days 1, 8, 15 and 22) or 20 mg in patients > 75 years old, Q4W. Dose level 3
* Belantamab-Mafodotin 2.5 mg/kg on day 1, every 4 weeks (Q8W)
* Carfilzomib 20/70 mg/m2 on days 1, 8, and 15, Q4W.
* Dexamethasone 40 mg weekly (days 1, 8, 15 and 22) or 20 mg in patients > 75 years old., Q4W

The rules applied for the Lead-in phase are as follows:

1. An initial cohort of 3 subjects is enrolled at the first dose level (DL1).
2. If 1/3 subjects develop a DLT, 3 additional patients will be included at the same dose level (DL1)
3. If 0/3 subjects develop a DLT, 3 additional patients will be included at the next dose level (DL2, dose level 2).
4. If 1/3 subjects develop a DLT, 3 additional patients will be included at the same dose level (DL2, dose level 2).
5. If 0 of the 3 new subjects develops a DLT (for a total of 0-1/6 patients with a DLT at this dose level), 3 new subjects will be included in DL3 (dose level 3).
6. If 1 of the 3 new subjects develops a DLT (for a total of 0-1/6 patients with a DLT at this dose level), 3 new subjects will be included at the same dose level (DL3, dose level 3)
7. If 0 out of the 3 new subjects develops a DLT, 3 additional subjects will be included in the same dose level. If 0-1 out of 6 patients developed a DLT, this dose will be considered the maximum tolerated dose (MTD) and will be explored in the expansion phase (phase 2).
8. If ≥2/3 subjects develop a DLT, dose level will be de-escalated (previous dose level) with the same rules as described above.

Dose limiting toxicities (DLTs) will be evaluated during the DLT evaluation period. The DLT evaluation period will be defined as the first 4-weeks treatment cycle for each cohort.

Patients participating in the Lead-In-Phase must undergo a complete ophthalmologic examination at the end of the DLT evaluation period (4-weeks) and before starting Cycle 2.

Subjects will be considered evaluable for the assessment of DLT if they:

* Received at least 1 dose of belantamab mafodotin + Kd and experience a DLT, OR
* Received at least 1 dose of belantamab mafodotin, 3 doses of Carfilzomib and 3 doses of Dexamethasone and complete the safety follow-up through the end of the DLT evaluation period.

Non-evaluable subjects will be replaced.

Phase 2 (Expansion Phase, n= up to 60 patients)

Combination treatment will be administered at the RP2D based on the results of the phase 1 dose escalation part of the study:

* Belantamab mafodotin on day 1 at the RP2D, every 8 weeks, intravenously (IV).
* Carfilzomib will be given at the RP2D weekly IV on days: 1, 8, and 15 of every 4-week cycle (Q4W).
* Dexamethasone will be given at the dose of 40 mg (or 20 mg if patient > 75 years old) on days: 1, 8, 15 and 22 Q4W.

From month 13 onwards carfilzomib treatment will be given on day 1 and 15 of every 4-weeks cycles. Belantamab will be given at the RP2D every 8 weeks and Dexamethasone 40mg on days 1, 8, and 15 of every 4-week cycle.

The trial has the following objectives:

Primary objectives (PO):

Phase 1 PO1: To determine the maximum tolerated dose, and the recommended phase 2 dose of belantamab mafodotin in combination with carfilzomib and dexamethasone.

Phase 2 PO2: To evaluate the efficacy in terms of complete response rate and rates of minimal residual negativity after 12 months of therapy with belantamab mafodotin combined with carfilzomib and dexamethasone.

PO3: To evaluate safety and tolerability of the combination of belantamab mafodotin plus carfilzomib and dexamethasone.

Secondary Objectives (SO):

SO1: To determine time to event data of the combinations: Progression-free survival, progression-free survival at 12 months, duration of response, time to response, and overall survival.

SO2: Evaluate deepening of response during continuous therapy at 12, and 24 months.

SO3: Evaluate sustained MRD rate at 1 and 2 years. SO4: Evaluate the rate of conversion from MRD positivity to MRD negativity during the treatment (yearly).

SO5: To assess the safety of the combination of belantamab mafodotin + Kd, as well as the incidence of corneal and ophthalmologic adverse events.

ELIGIBILITY:
Inclusion Criteria:

Participant must be able to understand the study procedures

1. Patient is, in the investigator's opinion, willing and able to comply with the protocol requirements.
2. Patient has given voluntary written informed consent before performance of any study-related procedure nor part of normal medical care, with the understanding that consent may be withdrawn by the patient at any time without prejudice to their future medical care.
3. Relapse multiple myeloma patients that have received at least 1 and no more than 3 prior lines of therapy. Induction, intensification with high-dose melphalan and stem cell transplant and maintenance is considered one line of treatment.
4. Patients must be refractory to lenalidomide. Refractoriness is defined as progression while receiving lenalidomide or in the first 60 days after the last dose of lenalidomide.

   Refractoriness would be defined regardless of the dose of lenalidomide received, and the schedule or whether it was given alone or in combination.
5. Patients can have received prior treatment with proteasome inhibitors. Patients with prior bortezomib treatment are eligible regardless of refractory status. Prior carfilzomib treatment is allowed, provided that the patients achieve at least a partial response to prior carfilzomib, and that there is a treatment free interval of at least 6 months.
6. Participant must have a measurable secretory disease defined as either serum monoclonal protein of ≥ 0,5 g/dl or urine monoclonal (light chain) protein ≥ 200 mg/24 h. For patients whose disease is only measurable by serum FLC, the involved FLC should be ≥ 10mg/L (100 mg/dl), with an abnormal serum FLC ratio.
7. Participant must have an Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 2
8. Participant must be ≥ 18 years of age
9. Participant must have adequate organ function. Laboratory values that define adequate organ function for inclusion in study are as follow:

   HEMATOLOGIC Absolute neutrophil count (ANC) ≥1.5 X 109/L Hemoglobin ≥8.0 g/dL (prior red blood cell (RBC) transfusion or recombinant human erythropoietin use is permitted) Platelets ≥75 x 109/L for subjects in whom <50% of bone marrow nucleated cells are plasma cells; otherwise platelet count >50 × 10*9/L (prior platelet transfusion is permitted up to 7 days before the screening phase) Calcium corrected serum calcium <14 mg/dL (<3.5 mmol/L); or free ionized calcium <6.5 mg/dL (<1.6 mmol/L); HEPATIC Total bilirubin ≤1.5X ULN (Isolated bilirubin ≥1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%) ALT ≤2.5 X ULN AST ≤2.5 X ULN

   RENAL eGFRa ≥40 mL/min/ 1.73 m2 Spot urine (albumin/creatinine ratios) <500 mg/g (56 mg/mmol) OR Negative/trace (if ≥1+ only eligible if confirmed ≥ 500 mg/g (56 mg/mmol) by albumin/creatinine ratio (spot urine from first void) Urine Dipstick

   CARDIAC LVEF (echo) ≥ 40%
10. Female participants: contraceptive use should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies. A female participant is eligible to participate if she is not pregnant or breastfeeding, and at least one of the following conditions applies:

    * Is not a woman of childbearing potential (WOCBP) OR
    * Is a WOCBP and using a contraceptive method that is highly effective (with a failure rate of <1% per year), preferably with low user dependency, during the intervention period and for at least 4 months after the last dose of study intervention and agrees not to donate eggs (ova, oocytes) for the purpose of reproduction during this period. The investigator should evaluate the effectiveness of the contraceptive method in relationship to the first dose of study intervention.

    A WOCBP must have a negative highly sensitive serum pregnancy test (as required by local regulations) within 72 hours before the first dose of study intervention.

    The investigator is responsible for review of medical history, menstrual history, and recent sexual activity to decrease the risk for inclusion of a woman with a nearly undetected pregnancy.

    Nonchildbearing potential is defined as follows (by other than medical reasons):
    * ≥45 years of age and has not had menses for >1 year
    * Patients who have been amenorrhoeic for >2 years without history of a hysterectomy and oophorectomy must have a follicle stimulating hormone value in the postmenopausal range upon screening evaluation
    * Post-hysterectomy, post-bilateral oophorectomy, or post-tubal ligation.Documented hysterectomy or oophorectomy must be confirmed with medical records of the actual procedure or confirmed by an ultrasound. Tubal ligation must be confirmed with medical records of the actual procedure.
11. Male participants: contraceptive use should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.

    Male participants are eligible to participate if they agree to the following from the time of first dose of study until 6 months after the last dose of belantamab mafodotin to allow for clearance of any altered sperm:

    - Refrain from donating sperm

    PLUS either:
    * Be abstinent from heterosexual intercourse as their preferred and usual lifestyle (abstinent on a long term and persistent basis) and agree to remain abstinent OR
    * Must agree to use contraception/barrier as detailed below:

      * Agree to use a male condom, even if they have undergone a successful vasectomy and female partner to use an additional highly effective contraceptive method with a failure rate of <1% per year when having sexual intercourse with a WOCBP (including pregnant females).
12. All prior treatment-related toxicities (defined by National Cancer Institute- Common Toxicity Criteria for Adverse Events (NCI-CTCAE), version 4.0 must be ≤ Grade 1 at the time of enrolment except for alopecia
13. Participant must be able to understand the study procedures and agree to participate in the study by providing written informed consent

Exclusion Criteria:

1. Participant has a diagnosis of primary amyloidosis, monoclonal gammopathy of undetermined significance (MGUS), smoldering multiple myeloma (SMM), plasma cell leukemia or active POEMS syndrome at the time of screening.
2. Participant has invasive malignancies other than disease under study, unless the second malignancy has been medically stable for at least 2 years and, in the opinion of the principal investigators, will not affect the evaluation of the effects of clinical trial treatments on the currently targeted malignancy. Participants with curatively treated non-melanoma skin cancer may be enrolled without a 2-year restriction.
3. Participant has meningeal involvement of multiple myeloma.
4. Pregnant or breastfeeding females.
5. Participant is simultaneously enrolled in other interventional clinical trial.
6. Participant has used a systemic anti-myeloma drug within 14 days or five half-lives, whichever is shorter, preceding the first dose of study drug.
7. Participant has used an investigational drug within 14 days or five half-lives, whichever is shorter, preceding the first dose of study drug.
8. Prior treatment with a monoclonal antibody within 30 days of receiving the first dose of study drug.
9. Participant has received prior treatment with anti-BCMA agents.
10. Received plasmapheresis within 7 days prior to the first dose of study drug.
11. Participant has received prior radiotherapy within 2 weeks of start of study therapy.

    Participants must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis. A 1-week washout is permitted for palliative radiation (≤2 weeks of radiotherapy) to non-central nervous system (CNS) disease.
12. Participant has a known immediate or delayed hypersensitivity reaction or idiosyncratic reactions to belantamab mafodotin or drugs chemically related to belantamab mafodotin, or any of the components of the study treatment.
13. Participant has a known immediate or delayed hypersensitivity reaction or idiosyncrasy to other molecular antibodies.
14. Major surgery (except kyphoplasty) ≤ 4 weeks prior to initiating protocol therapy.
15. Participant has current corneal epithelial disease except mild changes in corneal epithelium
16. Participant has peripheral neuropathy or neuropathic pain grade ≥2, as defined by the National Cancer Institute Terminology Criteria for Adverse Events (NCI CTCAE) Version 4.0.
17. Participant evidence of cardiovascular risk including any of the following:

    * QTcF interval QTcF > 480 msec (the QT interval values must be corrected for heart rate by Fridericia's formula [QTcF])
    * Evidence of current clinically significant uncontrolled arrhythmias, including clinically significant ECG abnormalities such as 2nd degree (Type II) or 3rd degree atrioventricular (AV) block.
    * History of myocardial infarction, acute coronary syndromes (including unstable angina), coronary angioplasty, or stenting or bypass grafting within six months of Screening.
    * Class III or IV heart failure as defined by the New York Heart Association functional classification system [NYHA, 1994]
    * Uncontrolled hypertension, defined as an average systolic blood pressure ≥ 160 mmHg or diastolic ≥ 100 mmHg despite optimal treatment.
18. Participant has current unstable liver or biliary disease defined by the presence of ascites, encephalopathy, coagulopathy, hypoalbuminemia, esophageal or gastric varices, persistent jaundice, or cirrhosis. Note: Stable chronic liver disease (including Gilbert's syndrome or asymptomatic gallstones) or hepatobiliary involvement of malignancy is acceptable if otherwise meets entry criteria.
19. Presence of active renal condition (infection, requirement for dialysis or any other condition that could affect patient's safety). Participants with isolated proteinuria resulting from MM are eligible, provided they fulfil inclusion criteria.
20. Evidence of active mucosal or internal bleeding.
21. Use of contact lenses while participating in this study.
22. Any serious medical condition or psychiatric illness that would interfere in understanding of the informed consent form.
23. Uncontrolled endocrine diseases (i.e. diabetes mellitus, hypothyroidism or hyperthyroidism) (i.e. requiring relevant changes in medication within the last month, or hospital admission within the last 3 months).
24. Patients with acute diffuse infiltrative pulmonary disease and/or pericardial disease.
25. Patients with severe chronic obstructive pulmonary disease (COPD) or asthma with forced expiratory volume in the first minute (FEV1) less than 50%.
26. History of interstitial lung disease or ongoing interstitial lung disease. aa. Participant has an active infection requiring antibiotic, antiviral, or antifungal treatment bb. Participant has known HIV infection cc. Participant has presence of hepatitis B surface antigen (HBsAg), or hepatitis B core antibody (HBcAb at screening or within 3 months prior to first dose of study treatment.

dd. Participant has positive hepatitis C antibody test result or positive hepatitis C RNA test result at screening or within 3 months prior to first dose of study treatment.

Note: Participants with positive Hepatitis C antibody due to prior resolved disease can be enrolled, only if a confirmatory negative Hepatitis C RNA test is obtained.

Note: Hepatitis RNA testing is optional and participants with negative Hepatitis C antibody test are not required to also undergo Hepatitis C RNA testing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-12-20 (Actual); Primary Completion 2024-05 (Estimated); Study Completion 2028-05-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events (AEs) during the triplet-therapy in phase I. | At the end of the first 4-week cycle following a 3+3 design.
  To determine the maximum tolerated dose, and the recommended phase 2 dose of belantamab mafodotin in combination with carfilzomib and dexamethasone, number of participants with adverse events (AEs) during the triplet-therapy in phase 1 will be evaluated.
Overall Response Rate (ORR) | 12 months.
  Percentage of participants with a confirmed partial response (PR) or better (PR, VGPR, CR, sCR).
Minimal Residual Disease (MRD) negativity rate | At the time of CR/VGPR, and in all patients at month 12, 18, and 24, and yearly thereafter.
  The percentage of participants who are MRD negative by next-generation flow cytometry (NGF).
Complete Response Rate (CRR) | 12 months.
  The percentage of participants with a confirmed complete response (CR) or better (stringent complete response (CR, sCR)).
Incidence of deaths and primary cause of death. | Throughout the study. Approximately 60 months.
  Frequency and percentage of deaths and primary cause of death.
Incidence of adverse events (AEs). | Throughout the study. Approximately 60 months.
  Frequency and percentage of AEs
% of patients with changes in hematologic laboratory parameters | Throughout the study. Approximately 60 months.
  Percentage of patients who present differences in hematologic laboratory parameters from baseline values .
% of patients with changes in blood chemistry laboratory parameters | Throughout the study. Approximately 60 months.
  Percentage of patients who present differences in blood chemistry panel from baseline values.
Frequency of ocular findings on ophthalmic exam | Throughout the study. Approximately 60 months.
  Ocular findings on ophthalmic exam

SECONDARY OUTCOMES:
Duration of Response (DoR) | Throughout the study. Approximately 60 months.
  Time from first documented evidence of PR or better until progressive disease (PD) or death due to PD among participants who achieved PR or better.
Progression-Free Survival (PFS) | Throughout the study. Approximately 60 months.
  Time from the start of treatment until the earliest date of documented disease progression or death due to any cause.
Progression-Free Survival (PFS) at 12 months. | 12 months
  Time from the start of treatment until the earliest date of documented disease progression or death due to any cause.
Time to Response (TTR) | Throughout the study. Approximately 60 months.
  Time from the start of treatment and the first documented evidence of response (PR or better) among participants who achieve confirmed PR or better.
Overall Survival (OS) | Throughout the study. Approximately 60 months.
  Time from the start of treatment until the date of death due to any cause
Percentage of patients upgrading the response category | At 12 and 24 months
  Percentage of patients upgrading/deepening the response (converting from partial response to VGPR, etc.)
Percentage of patients achieving minimal residual disease negativity using EuroFlow Panel with a sensitivity of 10*(-6). | At 12, 18 and 24 months
  Percentage of patients achieving minimal residual disease negativity using EuroFlow Panel with a sensitivity of 10*(-6)
Percentage of patients converting from positive MRD to undetectable MRD following EuroFlow panel with a sensitivity of 10*(-6) | At 12, 24, 36, 48 and 60 months.
  Percentage of patients converting from positive MRD to undetectable MRD following EuroFlow panel with a sensitivity of 10-6
Incidence of Treatment related adverse events | Throughout the study. Approximately 60 months.
  Frequency and percentage of Treatment related adverse events
Percentage of patients discontinuing therapy due to AEs. | Throughout the study. Approximately 60 months.
  Percentage of patients discontinuing therapy due to AEs.
Percentage of patients requiring dose modifications. | Throughout the study. Approximately 60 months.
  Percentage of patients requiring dose modifications.

CONTACTS AND LOCATIONS:
Overall Officials: Paula Rodríguez Otero, Study Chair — Clínica Universidad de Navarra; María-Victoria Mateos, Study Chair — University of Salamanca; Jesús San Miguel Izquierdo, Study Chair — Clínica Universidad de Navarra
Locations (15):
- Spain (15):
  - Hospital Germans Trias i Pujol (ICO BADALONA), Badalona
  - Hospital Clinic, Barcelona
  - ICO Hospitalet, Bellvitge
  - H. Gregorio Marañón, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - H. Morales Meseguer, Murcia
  - HUCA, Oviedo
  - H. Son Llatzer, Palma de Mallorca
  - Clínica Universidad de Navarra (CUN), Pamplona
  - Hospital Universitario de Salamanca, Salamanca
  - H. Universitario de Canarias, Santa Cruz de Tenerife
  - H. Universitario Marqués de Valdecilla, Santander
  - Complejo Hospitalario Santiago (CHUS), Santiago de Compostela
  - Complejo Hospitalario Virgen del Rocío, Seville
  - H.U. La Fe, Valencia

REFERENCES:
- [Background] Berenson JR, Cartmell A, Bessudo A, Lyons RM, Harb W, Tzachanis D, Agajanian R, Boccia R, Coleman M, Moss RA, Rifkin RM, Patel P, Dixon S, Ou Y, Anderl J, Aggarwal S, Berdeja JG. CHAMPION-1: a phase 1/2 study of once-weekly carfilzomib and dexamethasone for relapsed or refractory multiple myeloma. Blood. 2016 Jun 30;127(26):3360-8. doi: 10.1182/blood-2015-11-683854. Epub 2016 May 12. PMID 27207788
- [Background] Chari A, Martinez-Lopez J, Mateos MV, Blade J, Benboubker L, Oriol A, Arnulf B, Rodriguez-Otero P, Pineiro L, Jakubowiak A, de Boer C, Wang J, Clemens PL, Ukropec J, Schecter J, Lonial S, Moreau P. Daratumumab plus carfilzomib and dexamethasone in patients with relapsed or refractory multiple myeloma. Blood. 2019 Aug 1;134(5):421-431. doi: 10.1182/blood.2019000722. Epub 2019 May 21. PMID 31113777
- [Background] Cowan AJ, Allen C, Barac A, Basaleem H, Bensenor I, Curado MP, Foreman K, Gupta R, Harvey J, Hosgood HD, Jakovljevic M, Khader Y, Linn S, Lad D, Mantovani L, Nong VM, Mokdad A, Naghavi M, Postma M, Roshandel G, Shackelford K, Sisay M, Nguyen CT, Tran TT, Xuan BT, Ukwaja KN, Vollset SE, Weiderpass E, Libby EN, Fitzmaurice C. Global Burden of Multiple Myeloma: A Systematic Analysis for the Global Burden of Disease Study 2016. JAMA Oncol. 2018 Sep 1;4(9):1221-1227. doi: 10.1001/jamaoncol.2018.2128. PMID 29800065
- [Background] Dimopoulos MA, Moreau P, Palumbo A, Joshua D, Pour L, Hajek R, Facon T, Ludwig H, Oriol A, Goldschmidt H, Rosinol L, Straub J, Suvorov A, Araujo C, Rimashevskaya E, Pika T, Gaidano G, Weisel K, Goranova-Marinova V, Schwarer A, Minuk L, Masszi T, Karamanesht I, Offidani M, Hungria V, Spencer A, Orlowski RZ, Gillenwater HH, Mohamed N, Feng S, Chng WJ; ENDEAVOR Investigators. Carfilzomib and dexamethasone versus bortezomib and dexamethasone for patients with relapsed or refractory multiple myeloma (ENDEAVOR): a randomised, phase 3, open-label, multicentre study. Lancet Oncol. 2016 Jan;17(1):27-38. doi: 10.1016/S1470-2045(15)00464-7. Epub 2015 Dec 5. PMID 26671818
- [Background] Lonial S, Lee HC, Badros A, Trudel S, Nooka AK, Chari A, Abdallah AO, Callander N, Lendvai N, Sborov D, Suvannasankha A, Weisel K, Karlin L, Libby E, Arnulf B, Facon T, Hulin C, Kortum KM, Rodriguez-Otero P, Usmani SZ, Hari P, Baz R, Quach H, Moreau P, Voorhees PM, Gupta I, Hoos A, Zhi E, Baron J, Piontek T, Lewis E, Jewell RC, Dettman EJ, Popat R, Esposti SD, Opalinska J, Richardson P, Cohen AD. Belantamab mafodotin for relapsed or refractory multiple myeloma (DREAMM-2): a two-arm, randomised, open-label, phase 2 study. Lancet Oncol. 2020 Feb;21(2):207-221. doi: 10.1016/S1470-2045(19)30788-0. Epub 2019 Dec 16. PMID 31859245
- [Background] O'Connor OA, Stewart AK, Vallone M, Molineaux CJ, Kunkel LA, Gerecitano JF, Orlowski RZ. A phase 1 dose escalation study of the safety and pharmacokinetics of the novel proteasome inhibitor carfilzomib (PR-171) in patients with hematologic malignancies. Clin Cancer Res. 2009 Nov 15;15(22):7085-91. doi: 10.1158/1078-0432.CCR-09-0822. Epub 2009 Nov 10. PMID 19903785
- [Background] Siegel DS, Martin T, Wang M, Vij R, Jakubowiak AJ, Lonial S, Trudel S, Kukreti V, Bahlis N, Alsina M, Chanan-Khan A, Buadi F, Reu FJ, Somlo G, Zonder J, Song K, Stewart AK, Stadtmauer E, Kunkel L, Wear S, Wong AF, Orlowski RZ, Jagannath S. A phase 2 study of single-agent carfilzomib (PX-171-003-A1) in patients with relapsed and refractory multiple myeloma. Blood. 2012 Oct 4;120(14):2817-25. doi: 10.1182/blood-2012-05-425934. Epub 2012 Jul 25. PMID 22833546
- [Background] Trudel S, Lendvai N, Popat R, Voorhees PM, Reeves B, Libby EN, Richardson PG, Anderson LD Jr, Sutherland HJ, Yong K, Hoos A, Gorczyca MM, Lahiri S, He Z, Austin DJ, Opalinska JB, Cohen AD. Targeting B-cell maturation antigen with GSK2857916 antibody-drug conjugate in relapsed or refractory multiple myeloma (BMA117159): a dose escalation and expansion phase 1 trial. Lancet Oncol. 2018 Dec;19(12):1641-1653. doi: 10.1016/S1470-2045(18)30576-X. Epub 2018 Nov 12. PMID 30442502
- [Background] Trudel S, Lendvai N, Popat R, Voorhees PM, Reeves B, Libby EN, Richardson PG, Hoos A, Gupta I, Bragulat V, He Z, Opalinska JB, Cohen AD. Antibody-drug conjugate, GSK2857916, in relapsed/refractory multiple myeloma: an update on safety and efficacy from dose expansion phase I study. Blood Cancer J. 2019 Mar 20;9(4):37. doi: 10.1038/s41408-019-0196-6. PMID 30894515
- [Background] Vij R, Siegel DS, Jagannath S, Jakubowiak AJ, Stewart AK, McDonagh K, Bahlis N, Belch A, Kunkel LA, Wear S, Wong AF, Wang M. An open-label, single-arm, phase 2 study of single-agent carfilzomib in patients with relapsed and/or refractory multiple myeloma who have been previously treated with bortezomib. Br J Haematol. 2012 Sep;158(6):739-48. doi: 10.1111/j.1365-2141.2012.09232.x. Epub 2012 Jul 30. PMID 22845873